CLINICAL TRIAL: NCT00822757
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Immunogenicity of a Single Dose of the Lyophilized Formulation of Merck Staphylococcus Aureus Vaccine (V710) in Healthy Adults
Brief Title: Safety and Immunogenicity Study of V710 Lyophilized Formulation (V710-004)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V710-004; 2007_531
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Results first posted 2011-11-21 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
Keywords: study in healthy subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): V710
  Interventions: Biological: Comparator: V710
- 2 (Placebo Comparator): Placebo
  Interventions: Biological: Comparator: placebo

INTERVENTIONS:
Biological: Comparator: V710 — Single dose V710 (60 Mcg/0.5 mL) by intramuscular injection.
  Arms: 1
Biological: Comparator: placebo — Single dose of buffered saline placebo (0.5 mL) by intramuscular injection.
  Arms: 2

SUMMARY:
This study is being performed to evaluate a single 60 Mcg dose of lyophilized formulation of Merck Staphylococcus aureus vaccine (V710) in healthy subjects. This study is intended to provide necessary safety and immunogenicity data for the lyophilized formulation of V710 prior to its subsequent evaluation in patients at risk for developing serious S. aureus infections.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age
* Good physical health based upon medical history and physical examination
* Willing and able to participate in the entire study duration
* Female subject with a negative urine pregnancy test immediately prior to study vaccination

Exclusion Criteria:

* Chronic skin infections or a chronic skin condition (e.g. psoriasis)
* Serious S. aureus infection in the last 12 months
* Allergy to aluminum-containing substance taken in the body or to any other vaccine component
* Oral temperature equal to or greater than 100.4ºF (38.0ºC), within the past 2 days
* Participation in a prior V710 vaccine clinical study
* Participation in any other clinical study in the past 4 weeks, or during the 3-month study duration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-08; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Harro CD, Betts RF, Hartzel JS, Onorato MT, Lipka J, Smugar SS, Kartsonis NA. The immunogenicity and safety of different formulations of a novel Staphylococcus aureus vaccine (V710): results of two Phase I studies. Vaccine. 2012 Feb 21;30(9):1729-36. doi: 10.1016/j.vaccine.2011.12.045. Epub 2011 Dec 20. PMID 22192849

RESULTS

PARTICIPANT FLOW:
Groups:
- V710 (60 mcg) Lyophilized: V710 (60 mcg) single dose at baseline.
- Placebo: Saline placebo single dose at baseline.
Period: Overall Study
Arm/Group | V710 (60 mcg) Lyophilized | Placebo
Started | 41 | 10
Completed | 41 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V710 (60 mcg) Lyophilized | Placebo | Total
Number analyzed (Participants) | 41 | 10 | 51
Age, Customized [Number; unit: participants]
  17 years of age and under | 0 | 0 | 0
  18 to 29 years of age | 6 | 1 | 7
  30 to 39 years of age | 5 | 0 | 5
  40 to 49 years of age | 8 | 4 | 12
  50 to 59 years of age | 1 | 0 | 1
  60 to 69 years of age | 10 | 5 | 15
  70 to 80 years of age | 11 | 0 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 4 | 26
  Male | 19 | 6 | 25

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Fold-rise (GMFR) After the Administration of the Lyophilized Formulation of V710 (60 mcg).
Description: Participants whose geometric mean fold-rise (GMFR) in anti-0657n IgG was measured 14 days after a single dose of the lyophilized formulation of V710 (60 mcg) by a LUMINEX™ assay for IgG antibodies directly binding to the 0651nI S. aureus antigen. The calculation of GMFR is based on the ratio of IgG Titers (geometric mean concentrations in which the units of measure are µg/mL) prevaccination (pre)/14 days postvaccination (postvac).
Time Frame: Prevaccination to 14 days postvaccination
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V710 (60 mcg) Lyophilized | Placebo
Number analyzed (Participants) | 41 | 10
Ratio | 5.3 [3.8 to 7.2] | 1.0 [0.9 to 1.0]

2. Other Pre Specified Outcome: GMFR by Age
Description: Participants whose geometric mean fold-rise (GMFR) in anti-0657n IgG was measured among two age groups (18 to 59 years of age and 60 to 70 years of age)14 days after a single dose of the lyophilized formulation of V710 (60 Mcg) by a LUMINEX™ assay for IgG antibodies directly binding to the 0657nI S.aureus antigen. The calculation of GMFR is based on the ratio of IgG Titers (geometric mean concentrations in which the units of measure are µg/mL) pre/14 days postvac.
Time Frame: Prevaccination to 14 days postvaccination
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V710 (60 mcg) Lyophilized | Placebo
Number analyzed (Participants) | 41 | 10
Ratio
  Age <60 years | 4.0 [2.6 to 6.2] | 0.9 [0.8 to 1.0]
  Age ≥60 years | 6.8 [4.3 to 10.8] | 1.0 [0.9 to 1.1]

3. Other Pre Specified Outcome: GMFR in Antibody Concentration From Baseline
Description: An assessment of the kinetics of the immune response in the V710 group over time from baseline measurement and all postvaccination time points (Days 10, 14, 28, and 84). The calculation of GMFR is based on the ratio of IgG Titers (geometric mean concentrations in which the units of measure are µg/mL) pre/all (10, 14, 28, and 84) days postvac.
Time Frame: Prevaccination to Days 10, 14, 28, and 84 postvaccination
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V710 (60 mcg) Lyophilized | Placebo
Number analyzed (Participants) | 41 | 10
Ratio
  Day 10 | 3.6 [2.6 to 5.0] | 1.2 [0.7 to 2.2]
  Day 14 | 5.3 [3.8 to 7.2] | 1.0 [0.9 to 1.0]
  Day 28 | 6.9 [4.8 to 9.9] | 0.9 [0.8 to 1.0]
  Day 84 | 7.8 [5.5 to 11.2] | 0.9 [0.8 to 1.1]

ADVERSE EVENTS:
Time Frame: All clinical adverse experiences (AEs) were followed for 14 days postvaccination, injection-site AEs and oral temperature for 5 days postvaccination, and vaccine-related serious AEs and deaths for 84 days postvaccination (entire duration of the study)
Groups:
- V710 (60 mcg) Lyophilized: V710 (60 mcg)single dose at baseline.
Arm/Group | V710 (60 mcg) Lyophilized | Placebo
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/10
Other Adverse Events (participants affected / at risk) | 15/41 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V710 (60 mcg) Lyophilized (N=41) | Placebo (N=10)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 5 (5) | 1 (1)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No